CLINICAL TRIAL: NCT02840136
Title: Optimisation, Valorisation and Application of UPLC-MS/MS Based Monitoring of Antibiotic Concentrations in Sputum of Cystic Fibrosis Patients - Part 3: Non-blank Sputum Samples for Method Optimisation and Validation
Brief Title: LC-MS/MS Based Method Development for the Monitoring of Antibiotic Concentrations in Sputum of Cystic Fibrosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of staff
Sponsor: University Ghent (Other)
Collaborators: King Baudouin Foundation (Other); Belgische Vereniging voor Strijd tegen Mucoviscidose (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EC UZG 2015/1504; B670201526932 (Other: Belgian registration)
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Cystic Fibrosis
Keywords: Respiratory infection; Antibiotic therapy; LC-MS/MS; Sputum antibiotic concentrations
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections | interventions — Piperacillin, Tazobactam Drug Combination; Meropenem; Ceftazidime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard of care (Experimental): Sputum is collected from patients receiving standard of care therapy with IV piperacillin-tazobactam, ceftazidime or meropenem
  Interventions: Drug: Piperacillin-tazobactam combination product; Drug: Meropenem; Drug: Ceftazidime

INTERVENTIONS:
Drug: Piperacillin-tazobactam combination product
Drug: Meropenem
Drug: Ceftazidime

SUMMARY:
In this trial, various factors that may influence the antibiotic concentrations measured in the sputum of cystic fibrosis patients are studied.

A first factor is aerosol use. As cystic fibrosis patients often use aerosols, such as hypertonic saline, dilution of the antibiotics in sputum can be expected. The extent of this dilution is unknown and will be determined by comparing sputum samples collected before and after the use of an aerosol.

A second factor is the homogeneity of the antibiotics within one sputum sample. Multiple aliquots of the same sputum sample will be compared.

A third factor is the variability between several sputum samples collected during a drainage session. The antibiotic concentrations in 3 separate sputum samples will be compared.

The final goal is to standardise the sputum sample collection and processing of the samples to ensure a accurate concentration measurements in sputum.

DETAILED DESCRIPTION:
Antibiotic therapy is a cornerstone in the management of cystic fibrosis (CF). Nevertheless, little research focusses on the actual concentrations reached in the lung secretions of CF patients. As the pathogens causing the expedited decline in lung function primarily reside in the lung secretions, many physicians are now interested in these data. Therefore, the investigators have developed and validated a liquid chromatography tandem mass spectroscopy (UPLC-MS/MS) method to quantify the intravenous administered beta-lactam antibiotics ceftazidime, piperacillin and meropenem, as well as inhaled aztreonam in the sputum of CF patients. Besides having a validated analytical method, the sample collection and sample preparation needs to be standardised as the well to ensure an accurate concentration measurement.

In this trial, three factors which may cause a bias in the concentration measurements in sputum are studied using sputum from patients receiving therapy with one of the IV antibiotics.

A first factor is aerosol use. As cystic fibrosis patients often use aerosols, such as hypertonic saline, Ventolin or Pulmozyme, dilution of the antibiotics in sputum can be expected. Likely, the moments at which patients use aerosols will need to be considered when collection sputum for antibiotic concentration measurements. To investigate the extent and duration of a concentration change induced by aerosol use, a sputum sample is collected before aerosol use and right after completion of the aerosol as well as 30 min, 1h and 2h after completion of the aerosol, more samples are collected.

A second factor is the homogeneity of the antibiotics within one sputum sample. Sputum samples generally have a heterogeneous appearance. To investigate if the distribution of antibiotics is heterogeneous as well, the concentration of multiple aliquots of the same sputum sample will be compared. Five aliquots will be tested and the remaining sputum is homogenised and analysed as well.

A third factor is the variability between several sputum samples collected during a autogenous drainage session. A drainage session lead by a physiotherapist takes approximately 30 minutes and aims to loosen and remove the thick lung secretions as much as possible. It can be assumed that sputum spontaneously expectorated in a drainage session originates from different parts of the lung. To verify if the antibiotics are homogeneously or heterogeneously distributed in the lungs, sputum samples are collected in the beginning, middle and at the end of the drainage session. The antibiotic concentrations in the 3 separate sputum samples will be compared.

The data originating from these 3 tests will allow to standardise the time point of sample collection with respect to aerosol therapy and autogenous drainage as well as to evaluate if homogenisation of the collected samples is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patient
* Sputum production
* Inclusion after receiving at least 3 days of IV therapy with ceftazidime, piperacillin-tazobactam or meropenem

Exclusion Criteria:

- Inability to expectorate sputum

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Concentration changes induced by aerosol use | 2 h
  The antibiotic concentration changes in sputum induced by aerosol use are monitored over a period of 2 hours
Antibiotic distribution in single sputum sample | 0 h
  In a single sputum sample, the homogeneity of the antibiotic distribution is evaluated
Antibiotic concentration in subsequently collected samples from the same patient | 30 min
  Antibiotic concentrations are measured in sputum samples collected at the beginning, middle and end of a 30 minute autogenic drainage session

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data generated in this trial will be published in a peer reviewed international journal. This way, concentration measurements in individual patients will be made available to the scientific community.